CLINICAL TRIAL: NCT03493035
Title: A Case-control Study of Independent Predictors of Middle Cerebral Artery Aneurysm.
Brief Title: Risk Factors of Middle Cerebral Artery Aneurysm.
Acronym: MCAA
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Wojciech Kaspera, Principal Investigator, Medical University of Silesia
Other Study IDs: SilesianMUNch1
Record Dates: First submitted 2018-01-05; First posted 2018-04-10 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Middle Cerebral Artery Aneurysm
Keywords: Middle Cerebral Artery; Cerebral Aneurysm; Transcranial Color-Coded Sonography; Three-Dimensional Computed Tomography Angiography
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCA aneurysm group: All patients with unruptured MCA aneurysm diagnosed on three-dimensional computed tomography angiography (3D CTA) and transcranial color-coded sonography (TCCS) .
  Interventions: Diagnostic Test: Computed tomography angiography (3D CTA); Diagnostic Test: Transcranial color-coded sonography (TCCS)
- non-MCA aneurysm group: All patients with no evidence of intracranial pathologies on 3D CTA and diagnosed on transcranial color-coded sonography (TCCS).
  Interventions: Diagnostic Test: Computed tomography angiography (3D CTA); Diagnostic Test: Transcranial color-coded sonography (TCCS)

INTERVENTIONS:
Diagnostic Test: Computed tomography angiography (3D CTA) — CTA scans data in DICOM format was used to morphometric analysis of aneurysmal and non-aneurysmal MCA bifurcations.
Diagnostic Test: Transcranial color-coded sonography (TCCS) — TCCS was used to assess of hemodynamic parameters of aneurysmal and non-aneurysmal MCA bifurcations.

SUMMARY:
According to the current view, cerebral aneurysms are acquired degenerative lesions resulting from hemodynamic stress. This single-center case-control study will be carried out at the Department of Neurosurgery, Regional Hospital in Sosnowiec, Medical University of Silesia in Katowice, Poland between June 2015 and June 2017. The aim of the study is to determine morphometric and hemodynamic parameters of aneurysmal and non-aneurysmal middle cerebral artery (MCA) bifurcations and to analyze their relationship with aneurysm formation. A minimum of 75 cases and 75 age- and sex-matched controls will be required for the study. Characteristics of the MCA bifurcations will be determined with computed tomography angiography (CTA) and transcranial color-coded sonography (TCCS). The following variables will be evaluated as potential risk factors for MCA aneurysm formation: radii and cross-sectional area of the main MCA trunk and its branches, tortuosity of MCA trunk, asymmetry ratio, area ratio, the angle between the post-bifurcation branches, the angles between the MCA trunk and the larger and smaller branch, volume flow rate, mean flow velocity and pulsatility index of the MCA. All morphometric and hemodynamic parameters will be assessed as potential risk factors for MCA aneurysm formation.

DETAILED DESCRIPTION:
Current evidence suggests that a principal factor involved in formation, enlargement and rupture of cerebral aneurysms are hemodynamic forces acting at arterial bifurcation. The objective of this case-control study is to determine morphometric and hemodynamic parameters of aneurysmal and non-aneurysmal MCA bifurcations and to analyze their relationship with aneurysm formation. This single-center case-control study will be carried out at the Department of Neurosurgery, Regional Hospital in Sosnowiec, Medical University of Silesia in Katowice, Poland between June 2015 and June 2017. The study will include patients (cases) with unruptured MCA aneurysm diagnosed on three-dimensional computed tomography angiography (3D CTA). The controls will be patients with no evidence of intracranial pathologies on 3D CTA, referred to establish the etiology of minor symptoms, such as headache or vertigo. A minimum of 75 cases and 75 age- and sex-matched controls will be required for the study.

CTA scans data in DICOM format will be transferred to Mimics Innovation Suite (MIS) platform (Materialise, Leuven, Belgium). Image segmentation and creation of three-dimensional (3D) models will be carried out with Mimics v.17.0 MIS software (Materialise, Leuven, Belgium). The segmentation process will include main trunks of the MCA and the post-bifurcation branches. Trifurcations of the main MCA trunk will be excluded from the morphometric analysis. MCA bifurcations from the aneurysm patients will be divided into two groups: the An group with aneurysmal MCA bifurcations and the non-An group with contralateral non-aneurysmal MCA bifurcations. Also, MCA bifurcations from the controls will be divided into two groups: R-MCA group with bifurcations of the right MCA and the L-MCA group with bifurcations of the left MCA. Morphometric analysis will include the following parameters: radii and cross-sectional area of the main MCA trunk and its branches (for the larger and smaller branch, respectively), tortuosity of MCA trunk, asymmetry ratio, area ratio, the angle between the post-bifurcation branches, the angles between the MCA trunk and the larger and smaller branch. All TCCS examinations will be performed using a Vivid 3 Pro (GE Healthcare, Chicago, Illinois, USA) equipped with a multi-frequency transcranial probe (1.5-3.6 MHz). Angle-corrected mean blood flow velocity, peak systolic velocity and end-diastolic velocity will be measured for both MCAs. Pulsatility index and volume flow rate in each vessel will be calculated as well. The protocol of the study was approved by the Institutional Review Board, and written informed consent will be sought from all the study participants. All morphometric and hemodynamic parameters will be assessed as potential risk factors for MCA aneurysm formation.

ELIGIBILITY:
Definition and recruitment of cases The study will include patients (further referred to as cases) with unruptured MCA aneurysm diagnosed on three-dimensional computed tomography angiography (3D CTA).

Case inclusion criteria

* all patients with unruptured MCA aged between 18-75 years Case exclusion criteria
* refusal to participate in the study
* inability to give informed consent
* presence of multiple cerebral aneurysms
* presence of pathologies, other than MCA aneurysm, in the central nervous system that could have a potential effect on cerebral blood flow (e.g. ischemic stroke, intracerebral or subarachnoid hemorrhage)
* severe systemic disorders (e.g. neoplastic disease)
* severe heart failure or multi-organ failure
* hemodynamically significant internal carotid artery stenosis
* pregnancy
* family history of cerebral aneurysms.

Definition and recruitment of controls The controls will be patients with no evidence of intracranial pathologies on 3D CTA, referred to establish the etiology of minor symptoms, such as headache or vertigo.

Inclusion criteria for the controls

* all patients aged between 18-75 years with no evidence of intracranial pathologies on 3D CTA Exclusion criteria for the controls
* refusal to participate in the study
* inability to give informed consent
* presence of pathologies in the central nervous system that could have a potential effect on cerebral blood flow (e.g. ischemic stroke, intracerebral or subarachnoid hemorrhage)
* severe systemic disorders (e.g. neoplastic disease)
* severe heart failure or multi-organ failure
* hemodynamically significant internal carotid artery stenosis
* pregnancy
* family history of cerebral aneurysms.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients (further referred to as cases) with unruptured MCA aneurysm diagnosed on three-dimensional computed tomography angiography (3D CTA).
  The controls will be patients with no evidence of intracranial pathologies on 3D CTA, referred to establish the etiology of minor symptoms, such as headache or vertigo.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Computed tomography angiography (CTA) analysis of the cross-sectional area of the MCA bifurcations. | from 16 June 2015 to 15 June 2017
  CTA scans in DICOM format will be used to create three-dimensional (3D) models of MCA bifurcation using Mimics Innovation Suite platform (Materialise, Leuven, Belgium). The points including the largest curvature of MCA main trunk and two post-bifurcations branches will be automatically calculated according to the centreline fitted with a computer-aided design (CAD) tool. In these points the cross-sectional area (mm2) of the MCA trunk and its two post-bifurcation branches will be calculated automatically.
Computed tomography angiography (CTA) analysis of the best fit diameter of the MCA bifurcations. | from 16 June 2015 to 15 June 2017
  CTA scans in DICOM format will be used to create three-dimensional (3D) models of MCA bifurcation using Mimics Innovation Suite platform (Materialise, Leuven, Belgium). The points including the largest curvature of MCA main trunk and two post-bifurcations branches will be automatically calculated according to the centreline fitted with a computer-aided design (CAD) tool. In these points the best fit diameter (mm) of the MCA trunk and its two post-bifurcation branches will be calculated automatically.
Computed tomography angiography (CTA) analysis of the angles between the MCA bifurcations components. | from 16 June 2015 to 15 June 2017
  CTA scans in DICOM format will be used to create three-dimensional (3D) models of MCA bifurcation using Mimics Innovation Suite platform (Materialise, Leuven, Belgium). The points of the largest curvature of MCA main trunk and two post-bifurcations branches will be calculated according to the centreline fitted automatically with a computer-aided design (CAD) tool. The centrelines and the largest curvature points will be exported to 3-matic v.9.0 MIS software. Three points of the largest curvatures (the main MCA trunk and two post-bifurcations branches) together with the point of the intersection of both centrelines passing through the main trunk MCA and both branches will determine the arms and the apex of the three angles. The following angle values will be calculated automatically: the angle between the post-bifurcation branches (α angle) and the angles between the MCA trunk and the larger and the smaller branches (β and γ angle).
Pulsatility Index (PI) as calculated from transcranial color-coded sonography (TCCS) blood flow velocities (cm/s) | from 16 June 2015 to 15 June 2017
  The assessment of blood flow velocities in both MCAs will be performed by transcranial color-coded sonography (TCCS) using a Vivid 3 Pro (GE Healthcare, Chicago, Illinois, USA) equipped with a multi-frequency transcranial probe (1.5-3.6 MHz). For both MCAs the following will be automatically measured:
  1. mean blood flow velocity (V) [cm/s]
  2. peak systolic velocity (Vps) [cm/s]
  3. end-diastolic velocity (Ved) [cm/s] The velocity measurements will be used to calculate in each vessel the pulsatility index (PI), calculated using the following formula: PI=(Vps-Ved)/V
Volume Flow Rate (VFR) as calculated from transcranial color-coded sonography (TCCS) blood flow velocities (cm/s) | from 16 June 2015 to 15 June 2017
  The assessment of blood flow velocities in both MCAs will be performed by transcranial color-coded sonography (TCCS) using a Vivid 3 Pro (GE Healthcare, Chicago, Illinois, USA) equipped with a multi-frequency transcranial probe (1.5-3.6 MHz). For both MCAs the following will be automatically measured:
  1. mean blood flow velocity (V) [cm/s]
  2. peak systolic velocity (Vps) [cm/s]
  3. end-diastolic velocity (Ved) [cm/s] The velocity measurements will be used to calculate in each vessel the volume flow rate (VFR) using the following formula: VFR=V*p, where p - a cross-sectional area of the main MCA trunk, calculated from the morphometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Kaspera, MD, PhD, Principal Investigator — Medical University of Silesia
Locations (1):
- Wojciech Kaspera, Sosnowiec, Smorzykk@gmail.com, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available for 5 years after study completion.
Access Criteria: Data will be shared electronically by email or by depositing on a secure file share server depending on file type and size. If necessary, non-confidential files will be supplied on a data CD or USB flash drive. When requested, the data will be made available by the PI provided the request does not interfere with publication, compromise intellectual property interests, or precede data analysis. The data acquired and preserved will be governed by Medical University of Silesia policies regarding intellectual property, record retention, and data management.

REFERENCES:
- [Result] Ingebrigtsen T, Morgan MK, Faulder K, Ingebrigtsen L, Sparr T, Schirmer H. Bifurcation geometry and the presence of cerebral artery aneurysms. J Neurosurg. 2004 Jul;101(1):108-13. doi: 10.3171/jns.2004.101.1.0108. PMID 15255260
- [Result] Bor AS, Velthuis BK, Majoie CB, Rinkel GJ. Configuration of intracranial arteries and development of aneurysms: a follow-up study. Neurology. 2008 Feb 26;70(9):700-5. doi: 10.1212/01.wnl.0000302176.03551.35. PMID 18299521
- [Result] Rossitti S. Shear stress in cerebral arteries carrying saccular aneurysms. A preliminary study. Acta Radiol. 1998 Nov;39(6):711-7. doi: 10.3109/02841859809175503. PMID 9817048
- [Result] Kaspera W, Ladzinski P, Larysz P, Hebda A, Ptaszkiewicz K, Kopera M, Larysz D. Morphological, hemodynamic, and clinical independent risk factors for anterior communicating artery aneurysms. Stroke. 2014 Oct;45(10):2906-11. doi: 10.1161/STROKEAHA.114.006055. Epub 2014 Aug 28. PMID 25169949
- [Result] Tutuncu F, Schimansky S, Baharoglu MI, Gao B, Calnan D, Hippelheuser J, Safain MG, Lauric A, Malek AM. Widening of the basilar bifurcation angle: association with presence of intracranial aneurysm, age, and female sex. J Neurosurg. 2014 Dec;121(6):1401-10. doi: 10.3171/2014.8.JNS1447. Epub 2014 Oct 3. PMID 25280096
- [Result] Baharoglu MI, Lauric A, Safain MG, Hippelheuser J, Wu C, Malek AM. Widening and high inclination of the middle cerebral artery bifurcation are associated with presence of aneurysms. Stroke. 2014 Sep;45(9):2649-55. doi: 10.1161/STROKEAHA.114.005393. Epub 2014 Aug 12. PMID 25116869
- [Result] Can A, Ho AL, Dammers R, Dirven CM, Du R. Morphological parameters associated with middle cerebral artery aneurysms. Neurosurgery. 2015 Jun;76(6):721-6; discussion 726-7. doi: 10.1227/NEU.0000000000000713. PMID 25734323
- [Result] Sasaki T, Kakizawa Y, Yoshino M, Fujii Y, Yoroi I, Ichikawa Y, Horiuchi T, Hongo K. Numerical Analysis of Bifurcation Angles and Branch Patterns in Intracranial Aneurysm Formation. Neurosurgery. 2019 Jul 1;85(1):E31-E39. doi: 10.1093/neuros/nyy387. PMID 30137458

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03493035/Prot_SAP_000.pdf